CLINICAL TRIAL: NCT03939507
Title: A Prospective Study on Long-term Outcome and Potential Usefulness fo an Intervention Aimed at Reducing Adverse Effects in Patients With Refractory Epilepsy
Brief Title: Outcome Study in Refractory Epilepsy (SOPHIE)
Acronym: SOPHIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Collaborators: University of Catanzaro (Other); University of Bologna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FARM52K2WM_003
Record Dates: First submitted 2019-04-18; First posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Epilepsy
Keywords: epilepsy,; outcome; antiepileptic drugs; toxicity
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: In the randomized assessment, patients meeting eligibility were randomized to two groups. In the intervention group, AEP score results were made available to the treating physician at each assessment visit, while in the other group AEP scores were only made available at the end of follow-up.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): AEP score results were made available to the treating physician at each assessment visit.
  Interventions: Other: AEP score available to the treating physician
- Control group (No Intervention): AEP scores were only made available at the end of follow-up.

INTERVENTIONS:
Other: AEP score available to the treating physician — the treating physician knew the AEP score results
  Arms: Intervention group

SUMMARY:
Over 1 million people in the European Union (EU) suffer from chronic refractory epilepsy. Their quality of life (QoL) is severely affected by seizures and by the adverse effect of antiepileptic drug (AED) treatment. Several new AEDs have been introduced in recent years, but their impact on the long-term outcome in these patients has been inadequately explored. Preliminary data from the U.S. suggests that using a standardize toll to quantitate adverse AED effects can improve outcome, but the general applicability of these findings is unclear.

Objectives: 1) To assess prospectively AED utilization patterns in patients with refractory epilepsy ; 2) to assess how such treatments and other variables correlated with seizure control, adverse effects, and QoL in these patients; 3) to establish the impact of a standardized evaluation of adverse effects on clinical outcome.

Methods: The project included a core observational study and a randomized intervention in a subcohort.

In the core (observational) study, 1,000 consecutive refractory epilepsy patients were enrolled and followed-up prospectively at 10 centres in Italy. The following parameters were recorded at 0 (entry), 6, 12 and 18 months: (i) drug therapy; (ii) seizure frequency; (iii) adverse events based on medical examination and non-structured interview; (iii) treatment costs and, (iv) for patients above age 16, standardized questionnaires for adverse effects (AEP), depressive symptoms (Becks Depression Scale, BDS), QoL (QOLIE-31) and clinical global impression (CGI). The primary outcome (changes in QOLIE-31 scores) will be related to the other variables measured.

In the randomized intervention, the subcohort meeting specific eligibility criteria (age >16 years, no progressive disorder, AEP score>=45 ) was randomized to two groups. In the intervention group, AEP score results were made available to the physician at each visit, while in the other group AEP scores were only made available at the end of follow-up. Primary outcome were changes in AEP score.

DETAILED DESCRIPTION:
With a prevalence of about 0.8% in the general population, chronic active epilepsy is the most common serious neurological disorder and affects 3.7 million people in the EU alone. While the majority of patients with epilepsy can be fully controlled by available medications, about 40% fail to achieve seizure control. Refractory epilepsy is associated with poor quality of life (QoL), due to the consequences of seizures, the burden of adverse effects of antiepileptic drugs (AEDs), and associated comorbidities, especially depressed mood. In addition to human suffering, refractory epilepsy entails major costs: observational studies in Italy estimated an annual medical costs at 2,190 in adults, or 3,268 euros in children.

The study had a prospective design and mainly observational design (core study). A subgroup of patients, participated in a randomized assessment (controlled study) of the impact of utilizing a standardized tool for the assessment of adverse effects.

For the core study, the study population was represented by 1,000 consecutive consenting patients with refractory epilepsy seen as in- or outpatients at 10 major secondary/tertiary referral centres in Italy. "Refractory epilepsy" was defined as "the persistence of seizures after adequate attempts with the maximally tolerated dosage of one or more appropriate primary AEDs, excluding situations where a meaningful dose escalation was prevented by allergic or idiosyncratic adverse reactions" and at least one seizure during the previous 3 months while at steady state on the current treatment schedule. The degree of refractoriness was classified into categories.

A subcohort of patients included in the study took part in a randomized assessment of the usefulness of providing the treating physician with a standardized assessment of the adverse effect profile. The subcohort was represented by all patients enrolled in the core study who met at the first assessment visit the following additional eligibility criteria: (i) age >16 years; (ii) no progressive disorder; (iii) ability to complete the Adverse Profile AEP questionnaire, and (iv) an AEP score >=45.

For the core study, the approach was observational and the study did not interfere with clinical management. All patients were treated as considered best by the attending physician. Results of questionnaires were not made available to the treating physician until the end of the study, except for the AEP questionnaire data that were fed back to the physician only for a subgroup of patients included in the randomized assessment.

In the randomized assessment, patients meeting eligibility were randomized to two groups. In the intervention group, AEP score results were made available to the treating physician at each assessment visit, while in the other group AEP scores were only made available at the end of follow-up. Evaluations were identical to those carried out in the core study.

Except for making available the AEP scores to the treating physician, the procedures used for the collection and the handling of the information were identical in the core study and the randomized assessment. Patients were seen in the clinic at the following times: 0 (enrolment), 6, 12 and 18 months. At the first visit, detailed information were collected about demographics, medical history and current medical status. At this visit and at each of the other visits, the following information were collected:

* QOLIE-31 scores (only patients aged >16years), using the validated epilepsy-specific questionnaire, which is the most widely used for QoL tool in epilepsy in different countries;
* BDI scores (only patients aged >16years), using the validated inventory developed by Beck (1961), shown to have reliability and sensitivity in different settings, including refractory epilepsy ;
* AEP scores (only patients aged >16years), using the epilepsy-specific validated scale developed by prof. Baker ;
* A 5 digit Global Impression Scale for clinical change, compiled separately by the physician and by the patient/caregiver;
* Seizure frequency, by using seizure diaries compiled by patients and/or caregivers.
* Adverse effects, through general and neurological examination and non-structured interview;
* Drug treatment details (including, when available, serum AED levels), from the prescriber and patient's interview, and drug load scores as described by prof. Deckers;
* Items to be used for cost calculations, based on patient's records of laboratory tests, doctor's visits, specialist consultations, treatments, hospital admissions, and day-hospital days during follow up.

The study duration was 36 months.

ELIGIBILITY:
Core study:

Inclusion Criteria:

* an established diagnosis of epilepsy;
* drug refractoriness, defined as persistence of seizures after adequately applied treatment(s) with one or more appropriate AEDs at maximally tolerated doses, excluding treatments whereby idiosyncratic reactions prevented titration to usually effective dosages;
* at least one seizure during the previous 6 months while at steady state on the currently used AED regimen;
* written informed consent.

Exclusion Criteria:

- not seizures during the previous 6 months

Inclusion Criteria for a subgroup of patients, who took part in a randomized assessment:

* age >16 years;
* no progressive disorder;
* ability to complete the Adverse Profile AEP questionnaire;
* an AEP score >=45

Exclusion criteria:

* age <16 years;
* progressive disorder;
* inability to complete the Adverse Profile AEP questionnaire;
* an AEP score <45

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2006-11-06 (Actual); Primary Completion 2009-07-16 (Actual); Study Completion 2009-07-16 (Actual)

PRIMARY OUTCOMES:
Quality Of Life In Epilepsy (QOLIE)-31 global score | Month 18
  The change in QOLIE-31 global score (final visit vs initial visit). QOLIE-31 is a widely used epilepsy-specific questionnaire
Adverse Events Profiles (AEP) score | Month 18
  The change in AEP score (final visit vs initial visit). The epilepsy-specific validated scale was used. Higher values represent a worse outcome.

SECONDARY OUTCOMES:
Retention patients and AntiEpileptic Drugs (AEDs) added/substituted | month 6, 12, 18
  Retention of patients on each of the AEDs added/substituted
Percentage of patients seizure free on each of the AEDs added/substituted | month 6, 12
  Percentage of patients free achieving 6- and 12-month seizure remission on each of the AEDs added/substituted
Percentage of patients with 50% seizure reduction on each of the AEDs added/substituted | month 6
  Percentage of patients with 50% seizure reduction over 6 months (vs 3-month period before enrollment) on each of the AEDs added/substituted
Percentage of patients free from seizures | month 6, 12
  Percentage of patients free from seizures during the last 6 and 12 months of follow-up
Percentage of patients with 50% seizure reduction | month 6
  Percentage of patients with 50% seizure reduction (vs 3-month period before enrollment) during the last 6 months of follow-up
QOLIE-31 scores | month 6, 12, 18
  Changes in QOLIE-31 scores over time
Beck Depression Inventory (BDI) scores | month 6, 12, 18
  Changes in Beck Depression Inventory (BDI) scores over time. Higher values represent a worse outcome.
AEP scores | month 6, 12, 18
  Changes in Adverse Effect Profile (AEP) scores over time
Clinical Global Impression (CGI) scores | month 6, 12, 18
  Changes in CGI scores over time. CGI is a 5 digit global impression scale for clinical change, compiled separately by the physician and by the patient/caregiver.
Number of AEDs | month 6, 12, 18
  Number of AEDs changed/substituted over the follow-up period
Total drug load | month 6, 12, 18
  Changes in total drug load during follow-up. Drug loads, estimated as the sum of the prescribed daily dose (PDD)/defined daily dose (DDD) ratio for each AED included in the treatment regimen, where PDD is the prescribed daily dose and DDD is the defined daily dose, which corresponds to the assumed average maintenance daily dose of a drug used for its main indication.
Adverse effects | month 6, 12, 18
  Adverse effects, recorded over time, through general and neurological examination and non-structured interview.
Cost data | month 6, 12, 18
  Cost data are based on patient's records of laboratory tests, doctor's visits, specialist consultations treatments, hospital admissions and day-hospital days during follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Perucca, Prof, Study Director — Clinical Pharmacology Unit, University of Pavia
Locations (1):
- Clinical Pharmacology Unit, University of Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beghi E, Gatti G, Tonini C, Ben-Menachem E, Chadwick DW, Nikanorova M, Gromov SA, Smith PE, Specchio LM, Perucca E; BASE Study Group. Adjunctive therapy versus alternative monotherapy in patients with partial epilepsy failing on a single drug: a multicentre, randomised, pragmatic controlled trial. Epilepsy Res. 2003 Nov;57(1):1-13. doi: 10.1016/j.eplepsyres.2003.09.007. PMID 14706729
- [Background] Beghi E, Garattini L, Ricci E, Cornago D, Parazzini F; EPICOS Group. Direct cost of medical management of epilepsy among adults in Italy: a prospective cost-of-illness study (EPICOS). Epilepsia. 2004 Feb;45(2):171-8. doi: 10.1111/j.0013-9580.2004.14103.x. PMID 14738425
- [Background] Devinsky O, Vickrey BG, Cramer J, Perrine K, Hermann B, Meador K, Hays RD. Development of the quality of life in epilepsy inventory. Epilepsia. 1995 Nov;36(11):1089-104. doi: 10.1111/j.1528-1157.1995.tb00467.x. PMID 7588453
- [Background] Jannuzzi G, Cian P, Fattore C, Gatti G, Bartoli A, Monaco F, Perucca E. A multicenter randomized controlled trial on the clinical impact of therapeutic drug monitoring in patients with newly diagnosed epilepsy. The Italian TDM Study Group in Epilepsy. Epilepsia. 2000 Feb;41(2):222-30. doi: 10.1111/j.1528-1157.2000.tb00144.x. PMID 10691121
- [Background] Kwan P, Brodie MJ. Early identification of refractory epilepsy. N Engl J Med. 2000 Feb 3;342(5):314-9. doi: 10.1056/NEJM200002033420503. PMID 10660394
- [Background] Gilliam F. Optimizing health outcomes in active epilepsy. Neurology. 2002 Apr 23;58(8 Suppl 5):S9-20. doi: 10.1212/wnl.58.8_suppl_5.s9. PMID 11971128
- [Background] Perucca E. Marketed new antiepileptic drugs: are they better than old-generation agents? Ther Drug Monit. 2002 Feb;24(1):74-80. doi: 10.1097/00007691-200202000-00013. PMID 11805726
- [Background] Perucca E. An introduction to antiepileptic drugs. Epilepsia. 2005;46 Suppl 4:31-7. doi: 10.1111/j.1528-1167.2005.463007.x. PMID 15968807
- [Background] Gilliam FG, Fessler AJ, Baker G, Vahle V, Carter J, Attarian H. Systematic screening allows reduction of adverse antiepileptic drug effects: a randomized trial. Neurology. 2004 Jan 13;62(1):23-7. doi: 10.1212/wnl.62.1.23. PMID 14718691
- [Background] Johnson EK, Jones JE, Seidenberg M, Hermann BP. The relative impact of anxiety, depression, and clinical seizure features on health-related quality of life in epilepsy. Epilepsia. 2004 May;45(5):544-50. doi: 10.1111/j.0013-9580.2004.47003.x. PMID 15101836
- [Derived] Franco V, Canevini MP, De Sarro G, Fattore C, Fedele G, Galimberti CA, Gatti G, La Neve A, Rosati E, Specchio LM, Striano S, Tinuper P, Perucca E; SOPHIE Study Group. Does screening for adverse effects improve health outcomes in epilepsy? A randomized trial. Neurology. 2020 Jul 21;95(3):e239-e246. doi: 10.1212/WNL.0000000000009880. Epub 2020 Jun 29. PMID 32601123